CLINICAL TRIAL: NCT03156101
Title: A Clinical Study Evaluating the Safety and Efficacy of BinD19 Treatment in Relapse or Refractory Acute Lymphoblastic Leukemia and Lymphoma Subjects
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of BinD19 Treatment in R/R ALL and Lymphoma Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen BinDeBio Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017ZDYFY-BinD19
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Relapsed B-cell Acute Lymphoblastic Leukemia; Refractory B-cell Acute Lymphoblastic Leukemia; Relapsed／Refractory B-cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BinD19 (Experimental): BinD19 (autologous T cells transduced with CD19 TCR-ζ/4-1BB vector) administered as an IV infusion on days 0, 1 and 2 in the absence of disease progression or unacceptable toxicity. Minimum/maximum dose: 1x10^6/kg / 1x10^7/kg administered to patients with R/R B cell Acute Lymphoblastic Leukemia (ALL) or Lymphoma.
  Interventions: Biological: BinD19

INTERVENTIONS:
Biological: BinD19 — Autologous T cells purified from the peripheral blood mononuclear cells of subjects, transduced with TCR-ζ/4-1BB lentiviral vector, expanded in vitro and then frozen for future administration.

SUMMARY:
This is a single arm, open-label, uni-center, phase I/II study to determine the safety and efficacy of an experimental therapy called BinD19 cells in patients with B-cell acute lymphoblastic leukemia or lymphoma, who are chemo-refractory, relapsed after allogeneic SCT, or are otherwise ineligible for allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.
* CD19+ leukemia or lymphoma
* Not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor
* Follicular lymphoma, previously identified as CD19+:
* Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)
* ECOG result is 0, 1 or 2.
* With normal heart, liver and kidney functions.
* Negative serum antibody for EBV, CMV, HBV, HCV, HIV and syphilis.
* Negative in pregnancy test （female subject only).

Exclusion Criteria:

* ECOG result is 3, 4 or 5.
* Pregnant or lactating women
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* HIV infection
* Enrolled to other clinical study in the last 4 weeks.
* Subjects with systemic auto-immune disease or immunodeficiency.
* Subjects with CNS diseases.
* Subjects with secondary tumors.
* Subjects with tumor infiltration in liver, brain or GI tract.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events [Safety and Feasibility] | Study treatment until Week 24
  Occurrence of study related adverse events defined as NCI CTCAE 4.0 > grade 3 possibly, probably, or definitely related to study treatment.

SECONDARY OUTCOMES:
Overall Response [Efficacy] | 5 years
  Efficacy assessments for ALL were performed based on bone marrow and blood morphologic criteria and physical examination findings. Efficacy assessments for Lymphoma were based on tumor load, B cell number and immunoglobulins.

CONTACTS AND LOCATIONS:
Overall Officials: QIU SHI Zhuang, PhD, Study Director — Shenzhen BinDeBio Ltd.
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Li X, Liu Y, Zhang Z, Zhang X, Huang J, Li H, Li F, Zhang L, Li L, Wu X, Ma W, Sun Z, Yu H, Zhou Z, Feng X, Cui K, Li Z, Zhang H, Zeng Y, Wan X, Chen YH, Zhang M, Zhang Y. A Phase I clinical trial of chimeric antigen receptor-modified T cells in patients with relapsed and refractory lymphoma. Immunotherapy. 2020 Jul;12(10):681-696. doi: 10.2217/imt-2020-0022. Epub 2020 Jun 25. PMID 32580597